CLINICAL TRIAL: NCT06249607
Title: Impact Of Mindfulness Breathing Versus Storytelling On Non- Specific Insomnia In Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohammed Abubaker Rabiee, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MindfulnessBreathing,Insomnia
Record Dates: First submitted 2023-09-28; First posted 2024-02-08 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Insomnia; Sleep Disorder
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Sleep Wake Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A: combined sleep hygiene and storytelling (Experimental)
  Interventions: Other: storytelling; Other: Sleep hygiene
- Group B: combined sleep hygiene and mindfulness breathing exercise group (Experimental)
  Interventions: Other: Mindfulness breathing; Other: Sleep hygiene
- Group C: sleep hygiene group (Other)
  Interventions: Other: Sleep hygiene

INTERVENTIONS:
Other: storytelling — Storytelling android program: Subjects in group A or the storytelling group will be given headphones to listen to stories for 30 min (i.e., between 9 and 10 pm). While the subject listens to the story, a relative will present in a corner of the room to record when they fell asleep, the relative will present again in the room to record the time of falling asleep. The intervention will be done 7 nights a week for a period of 6 weeks.
  Arms: Group A: combined sleep hygiene and storytelling
Other: Mindfulness breathing — android program: Individuals in group B are instructed to "sit upright in a comfortable position with eyes closed," "focus on diaphragm movements while breathing in a slow, deep, relaxed manner," and to nonjudgmentally acknowledge and accept "unwanted thoughts, ideas or images" and "return attention to the diaphragmatic breathing. In this exercise, individuals are instructed to notice the physical sensations of breathing, both inhalations and exhalations, with a focus on the natural rate of respiration as opposed to forcibly controlling the breath. Duration: 5 minutes in duration per session, before sleep for 7 days a week for a total duration of 6 weeks
  Arms: Group B: combined sleep hygiene and mindfulness breathing exercise group
Other: Sleep hygiene — Subjects in all groups will receive tips about healthy sleep
  * Maintain a regular sleep routine.
  * Avoid daytime naps.
  * Don't stay in bed awake for more than 5-10 minutes.
  * Don't watch TV, use the computer, or read in bed.
  * Drink caffeinated drinks with caution.
  * Avoid inappropriate substances that interfere with sleep.
  * Clean fresh air.
  * Have a quiet, comfortable bedroom.

SUMMARY:
This study will be conducted to compare between effects of mindfulness breathing and storytelling on insomnia in the elderly.

DETAILED DESCRIPTION:
Sufficient sleep is essential for optimum health just a few of the numerous processes occurring during sleep include memory consolidation, clearance of brain metabolites, and restoration of nervous, immune, skeletal, and muscular systems. Despite the significance of adequate sleep, insufficient or disturbed sleep is extremely common. For instance, thirty percent of employed adults report obtaining 6 or fewer hours of sleep per night, approximately one-third of all adults report significant sleep complaints, and the two most common sleep disorders, insomnia and sleep-disordered breathing (SDB), each have prevalence rates exceeding 10% in the adult population. Unfortunately, current approaches to treatment are limited .

Story telling is another common soothing bedtime routine for children that uses pictures and writing. It is also a nursing intervention that can be implemented to comfort hospitalized children with acute illness and increase enthusiasm. Story telling is a recommended activity that enhances sleep duration in children. Furthermore, it is considered a positive bedtime routine, in addition to praying and brushing teeth, compared to maladaptive bedtime routine, such as watching television, playing with gadgets, and playing games with high-level activities .

ELIGIBILITY:
Inclusion Criteria:

* Patients who have non-specific insomnia for one month at least.
* Their ages > 65 years.
* Medically stable patients.
* Current complaint of poor SQ (score > 5 of the SQ scale)
* Body mass index ≤ 35 kg/m2.

Exclusion Criteria:

* Patients having a well-structured diagnosis of relevant brain illness or
* any disease directly affects sleep.
* Any patient with unstable medical condition
* History of chronic insomnia
* Indication of receiving treatments for depression and anxiety
* Hearing problem

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 93 (Actual)
Dates: Start 2024-01-05 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-05 (Actual)

PRIMARY OUTCOMES:
The Pittsburgh Sleep Quality Index | baseline
  Pittsburgh Sleep Quality Index (PSQI) as a valid tool was used to measure the patients' SQ. This instrument was comprised of seven domains, including quality of subjective sleep, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, daytime dysfunction, and use of medication for sleep over the previous month. The score of the domains ranged from 0 = "No difficulty" to 3 = "Severe difficulty". A total score > 5 was considered to be indicative of poor SQ. A global score between 0 and 21 was derived by summing up the seven subscale scores
Actigraphy | baseline
  Actigraph (Actiwatch Minimitter Company, INC - Sunriver, OR, USA) will be placed on the non-dominant wrist and activities will be monitored continuously and recorded at one minute intervals during wakefulness and sleep.
  The times of wakefulness and sleep will be determined individually through a diary kept by the volunteers, together with the times calculated by the actigraph monitor.
  The participants will keep the device for a period of 7 days before the first and the last training session. The device will be removed only at bath time and replaced to the wrist immediately after.
  The information will be collected by the device and recorded by a validated algorithm (Minimitter Company - USA®) and transferred to a closed technology software installed on a computer.
  After analysis of the exams, the data will be plotted on a spreadsheet for statistical treatment

CONTACTS AND LOCATIONS:
Overall Officials: mohamed abubakr rabiee, PhD, Principal Investigator — physical therapy
Locations (1):
- Naser specialized hospital, Cairo, Egypt

REFERENCES:
- See also: ABCs of SLEEPING: A review of the evidence behind pediatric sleep practice recommendations — https://pubmed.ncbi.nlm.nih.gov/26551999/